CLINICAL TRIAL: NCT02565004
Title: Clinical and Laboratory Analysis of Familial Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150204; 15-C-0204
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Cancer
Keywords: Genetic; Sample Collection; Natural History
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients who were enrolled on protocol 09-C-0079, or family members of patients who were enrolled on protocol 09-C-0079
- 2: Individuals found to harbor a germline APC promoter 1B variant not previously enrolled in Cohort l.

SUMMARY:
Background:

DNA makes up the instruction book for people s cells. Cancer is a disease caused by DNA changes that build up and affect cell function. Researchers want to learn more about what may cause cancer by testing the DNA of people with the disease and their family members.

Objective:

To find DNA changes that may be inherited and may cause or influence whether a person gets cancer. To study families with clusters of cancer to find out if there is a DNA mutation specific to certain cancers.

Eligibility:

People 18 years of age and older who:

Participated in the familial genetic part of NIH study 09-C-0079, a previous study or had family members enrolled in this study

Design:

Participants may have been screened in the previous study. They will give permission for researchers to use their data and their tissue or blood samples collected in the study.

Participants may give blood samples.

At each stage of testing, participants will meet with a genetics health care provider. The provider will explain the tests and answer questions.

If researchers find a DNA change that might increase the risk for cancer or other health issues, they will confirm this result in a testing lab. This will require a blood sample.

Participants personal DNA data and health information will be put in a database for research purposes.

DETAILED DESCRIPTION:
Background:

* This study is to continue the analysis begun on 09C0079 which was focused on identification of the genetic mutation associated with a new gastric polyposis syndrome, Gastric Adenocarcinoma and Proximal Polyposis of the Stomach (GAPPS).
* GAPPS is an autosomal dominant gastric polyposis syndrome that confers a substantial risk for gastric adenocarcinoma and has been found to be associated with germline point variants in APC promoter 1B.
* At this time, any non-gastric phenotype associated with GAPPS is unknown and is being explored using a phenotyping survey interview.

Objective

- To specifically investigate families with clusters of cancer to determine if there is a potential familial genetic mutation specific to a particular cancer and if present, to compare these genetic abnormalities with individuals from the same family without cancer.

Eligibility:

* Participants must meet one of the following:

  * Have been previously enrolled on the familial genetic analysis arm of NIH study 09-C-0079; OR
  * Be family members of patients previously enrolled on the familial genetic analysis arm of 09-C-0079; OR
  * Have a documented pathogenic germline APC promotor 1B variant from a CLIA approved laboratory.
* Participants must be 10 years of age or older

Design:

* This protocol was originally opened to continue same use of research that was approved under protocol 09-C-0079, to analyze the data for publication, and to provide participants with any results of clinical and analytic validity and clinical utility.
* In a subsequent amendment carriers of a germline APC promoter 1B variant will participate in a phenotyping assessment survey interview to assess the phenotype of Gastric Adenocarcinoma and Proximal Polypopsis of the Stomach (GAPPS).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must meet one of the following:

  * Have been previously enrolled on the familial genetic analysis arm of NIH study 09-C-0079; OR
  * Be family members of patients previously enrolled on the familial genetic analysis arm of 09-C-0079; OR
  * Have a documented pathogenic germline APC promotor 1B variant from a CLIA approved laboratory.
* Participants must be 10 years of age or older

EXCLUSION CRITERIA:

Inability to provide informed consent.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants or family members of participants previously enrolled on the familial genetic analysis arm of NIH study 09-C-0079 (must be 10 years old or older, may be pregnant)
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
investigate relationship of familial genetic mutation to a particular cancer | 1 year
  linkage analysis performed for familial clustering of malignant and pre-malignant disease in families

SECONDARY OUTCOMES:
To assess the phenotype of Gastric Adenocarcinoma and Proximal Polyposis of the Stomach (GAPPS) | 1-2 years
  Descriptive statistics such as median, mean and standard deviation will be calculated for all continuous quantitative variables, including age of diagnosis, frequency and duration of symptoms and medication dosage. Frequency data will be calculated for categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Calzone, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0204.html